CLINICAL TRIAL: NCT00513513
Title: A Phase II, Open Label Trial in Treatment na�ve, HIV 1 Infected Subjects Who Will Receive TMC114/Rtv as a Monotherapy
Brief Title: TMC114-C227: A Study to Evaluate the Effectiveness and Safety of TMC114 (Darunavir) With a Low Dose of Ritonavir as Monotherapy (no Other Anti-HIV Drugs Will be Given) in Patients Who Have Never Been Treated With Antiretrovirals (Anti-HIV Drugs) Previously
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment.
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR010612
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; TMC114; Protease inhibitor; Darunavir; Antiretroviral agents; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TMC114 (darunavir) / ritonavir

SUMMARY:
This is an open label study (no placebos are used; all patients will receive the true medication) to evaluate the effectiveness of TMC114/rtv in treatment naÃ-ve (never previously received anti-HIV drugs), HIV 1 infected patients.

DETAILED DESCRIPTION:
This is an open label (no placebo), uncontrolled (all patients will receive TMC114 with ritonavir at the same dose, trial to investigate the sustained anti-viral activity of TMC114/rtv monotherapy in 24 treatment naïve, HIV 1 infected patients over a period of 48 weeks.TMC114, 800 mg daily (2 tablets of 400 mg [F021]) will be given together with 1 capsule (100 mg) of ritonavir.Initially 11 subjects (Panel A, screening viral load between 10000 and 100000 copies/mL) will be included and followed for 8 weeks. If after 8 weeks of dosing at least 7 subjects virologically respond (viral load <400 copies/mL), 13 additional patients (Panel B) will be included. If no virologic failure is observed in at least 18 out of 24 patients who complete 8 weeks of dosing, the trial will continue as planned. In case more than 6 patients in Panel A and Panel B develop a virologic failure after 8 weeks of treatment, the trial will be stopped to conclude the treatment is not effective.The 13 additional patients enrolled in Panel B should have a screening viral load between 20000 and 500000 copies/mL. The CD4+ cell count in all 24 patients should be > 100 cells/µL at screening. The patient's medical condition, adverse events (side effects), study medication compliance, and laboratory evaluations for effectiveness and safety will be assessed at regular intervals. At the end of the 48 weeks treatment period patients will be followed for an additional 4 weeks to evaluate any side effects or laboratory abnormalities. Treatment with TMC114/rtv will be extended for all patients who continue to benefit after 48 weeks. 2 oral tablets of TMC114 400 mg will be administered once daily with 1 capsule (100mg) of ritonavir for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented HIV-1 infection
* For the first 11 subjects (Panel A), screening plasma HIV-1 viral load is =10000 copies/mL and <100000 copies/mL
* For the second set of 13 patients (Panel B), plasma HIV-1 viral load is =20000 copies/mL and <500000 copies/mL
* Patients with CD4+ cell count above 100 cells/µl
* Patients have voluntarily signed the ICF
* Patients can comply with the protocol requirements
* Patient's general medical condition, in the investigator's opinion, does not interfere with the assessments and the completion of the trial.

Exclusion Criteria:

* Presence of any currently active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV Infection 1993) with some exceptions
* Previous or current use of antiretroviral (ARVs/anti-HIV drugs) (including both investigational as well as commercially available ARVs indicated for the treatment of HIV-infection and ARVs for treatment of hepatitis B infection with anti-HIV activity (e.g., adefovir)
* Having one of protocol listed 1 PI, NRTI, or NNRTI resistance associated mutation at screening
* Patients with primary HIV infection
* Female patients of childbearing potential without use of effective non-hormonal birth control methods or not willing to continue practicing these birth control methods for at least 30 days after the end of the treatment period
* Any active clinically significant disease (e.g., abnormal heart function, pancreatitis, acute viral infection) or findings during screening of medical history or physical examination that are expected to compromise the patient's safety or outcome in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate sustained anti-viral activity of TMC114/rtv monotherapy in treatment naive, HIV 1 subjects defined by decrease of >1 log viral load (VL) at week 4, VL <400 copies/ml at week 8 and VL< 50 copies/ml at weeks 24 and 48.

SECONDARY OUTCOMES:
The secondary objectives are to evaluate safety and tolerability of TMC114/rtv over 48 weeks, to evaluate immunologic response, to evaluate the possible development of resistance and to monitor potential changes in body shape.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited